CLINICAL TRIAL: NCT01912053
Title: An Open-label, Multicenter, Phase II Trial, to Evaluate the Efficacy of Intra-hepatic Administration of Yttrium 90-labelled Microspheres (Therasphere®, Nordion) in Association With Intravenous Chemotherapy With Gemcitabine and Cisplatin for the Treatment of Intra-hepatic Cholangiocarcinoma, First Line.
Brief Title: Efficacy Study of Intra-hepatic Administration of Therasphere® in Association With Intravenous Chemotherapy to Treat Cholangiocarcinoma
Acronym: MispheC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Center Eugene Marquis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-EB-CHOL-Th; 2012-001213-16 (EudraCT Number); A121007-71 (Registry Identifier: French National Health)
Record Dates: First submitted 2013-07-17; First posted 2013-07-30 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-01

CONDITIONS: Cholangiocarcinoma
Keywords: Intra-hepatic Cholangiocarcinoma treatment
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Association; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Therasphere® (Experimental): Therasphere® in association with Gemcitabine and Cisplatin
  Interventions: Radiation: Therasphere® in association with Gemcitabine and Cisplatin

INTERVENTIONS:
Radiation: Therasphere® in association with Gemcitabine and Cisplatin — Therasphere® is a radioelement
  Other Names: 90-Yttrium theraspheres

SUMMARY:
The purpose of this study is to assess efficacy and tolerance of intra-hepatic administration of Yttrium 90-labelled microsphere (Theraspheres®, Nordion) in association with intravenous chemotherapy with Gemcitabin and Cisplatin for the treatment of intra-hepatic cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed intra-hepatic cholangiocarcinoma.
2. Measurable target of at least 2 cm diameter.
3. Healthy liver or cirrhosis CHILD < B8.
4. WHO-PS: 0-1.
5. Age ≥ 18 years.
6. Non-Metastatic disease in extra-hepatic (are permitted: local lymph nodes < 3 cm, less than 5 lung nodes < 11 mm).
7. Creatinine clearance (calculated with Cockcroft and Gault formula) ≥ 55 ml/min, polymorphonuclear neutrophils ≥ 1500 G/L, platelets ≥ 80 G/L, prothrombin ≥ 40% (INR ≤ 2.3), serum albumin ≥ 28 g/l, serum bilirubin ≤ 3 x LSN.
8. Pregnancy test: negative for women of childbearing potential.
9. Reliable contraception for a childbearing couple, men and woman must have an reliable contraception during the treatment and until 6 months following the end of the treatment by chemotherapy
10. Signed informed consent form.
11. Patient with national health insurance.

Exclusion Criteria:

1. Pancreas cancer or duodenum cancer invading the bile duct or ampullary cancer. Cholangiocarcinoma of the bile ducts: hilar, main duct, gallbladder.
2. Extra-hepatic metastasis (including local lymph nodes measuring > 30 mm).
3. Primary sclerosing cholangitis.
4. History of chemoembolization or radioembolization.
5. Cirrhose CHILD > B7
6. Portal vein trunk tumoral thrombosis
7. History of hepato-biliary neo adjuvant or palliative chemotherapy and/or radiotherapy.
8. Contra indication of Gemcitabine and/or Cisplatin.
9. Other invasive active cancer, excepting in situ cervical cancer and basocellular or spino cellular skin cancer treated adequately. Any history of cancer not considered as completely cured for at least one year.
10. Technical failure of the diagnostic arteriography.
11. Extra hepatic uptake on the pre-therapeutic scintigraphy not manageable with an arteriography.
12. Dosimetry study predicting lung exposure > 30 Gy.
13. Any unstable medical history (diabetes, hypertension …).
14. History of organ transplant.
15. Symptomatic grade 1 angina pectoris or grade ≥ 2 angina pectoris.
16. An evolutive neuropathy.
17. Patient who already has been involved in a clinical trial with drug intake, whether this drug was experimental or not, within 30 days before.
18. Pregnant patient or patient with breastfeeding.
19. Patient under administrative supervision.
20. Regular follow-up impossible for various reasons (psychological, familial, economical, and social).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Radiological response rate to the treatment with the association of chemotherapy and radioembolization | 3 months after radioembolization
  Evaluation according RECIST 1.1 criteria. Rate will be reassessed every 8 weeks

SECONDARY OUTCOMES:
Tolerance of intra-hepatic administration of Yttrium 90-labelled microspheres in association with intravenous chemotherapy with Gemcitabine and Cisplatin assessed according NCI/CTC AE version 4. | Up to 24 months
  Grade 3-4 toxicity appearance.Time between 1st treatment administration and date of 1st appearance of a grade 3-4 toxicity or date of last toxicities assessment in case no grade 3-4 toxicity
Tumor markers changes (CA19.9, CEA and AFP) | Up to 24 months
  Markers will be analysed every 8 weeks during treatment period and if applicable every 12 weeks after surgery
Radiological response rate by the CHOI criteria | Up to 24 months
  every 8 weeks and every 12 weeks after surgery if applicable
Change in metabolic activity measured by TEP | Change from baseline in metabolic activity 15 and 24 weeks after last treatment by microspheres
Changes of liver volume | Up to 24 months
  Every 8 weeks during treatment and every 12 weeks after surgery if applicable
Tumoral and non-tumoral dosimetric assessment of the liver | Up to 6 months
  Data obtained from SPECT/CT performed at each hepatic scintigraphy

CONTACTS AND LOCATIONS:
Overall Officials: Eveline Boucher, MD, Principal Investigator — Centre Eugene Marquis
Locations (7):
- France (7):
  - Hôpital Beaujon - Service de Chirurgie, Clichy
  - Hôpital Henri Mondor, Créteil
  - Hôpital saint-Eloi, Montpellier
  - CHU Nancy - Hôpital Brabois, Nancy
  - CHU- Hotel Dieu, Nantes
  - CHU Poitiers, Poitiers
  - Centre Eugene Marquis, Rennes